CLINICAL TRIAL: NCT04147585
Title: Effects of an Intermittent Reduced Calorie Diet on Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Assistant Professor of Medicine (Gastroenterology and Hepatology), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 53161
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Diet Modification
Keywords: IBD; Crohn's disease; Diet; Fasting; Intermittent Reduced Calorie Diet; CD; intermittent fasting; FMD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Fasting; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Three cycles of a 5-day Intermittent Reduced Calorie Diet
  Interventions: Other: Intermittent Reduced Calorie Diet (IRCD)
- Control Arm (No Intervention): Regular Diet

INTERVENTIONS:
Other: Intermittent Reduced Calorie Diet (IRCD) — Three cycles of a 5-day Intermittent Reduced Calorie Diet over three months.
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to see how an Intermittent Calorie Reduced Diet (IRCD) that mimics fasting (also known as a fasting mimicking diet, FMD) effects inflammation in patients with mild to moderate Crohn's disease (CD). The diet may allow users to receive the benefits of fasting while also being able to enjoy food (the ingredients of which are GRAS (generally recognized as safe) by the Food and Drug Administration (FDA). Research on dietary interventions and CD are very limited. Diets that mimick fasting have been studied with support of the National Institute of Health and published in leading journals. This research investigates whether markers of inflammation decrease and/or quality of life increases after five-day periods of the IRCD, and may provide rationale for its use to treat CD.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Crohn's disease (CDAI score 151-450)
* Between the ages of 18-70 (inclusive)

Exclusion Criteria:

* Women who are pregnant, nursing or expect to be pregnant
* Individuals allergic to nuts
* Individuals with a body mass index (BMI) lower than 18
* Individuals diagnosed with a serious medical condition (unless approved in writing by a physician)
* Individuals who have been severely weakened by a disease or medical procedure
* Individuals who are taking medication which may not be safely consumed with a calorie restricted diet
* Individuals with diabetes who are taking anti-diabetic drugs associated with risk of hypoglycemia
* Individuals with more than mild-moderate cardiovascular disease or life-threatening cancer (as determined by patient's physician) unless approved by a physician
* Individuals with history of severe cardiac disease (particularly uncompensated congestive heart failure NYHA grade 2 or more or LVEF < 40%)
* Individuals with a history of syncope
* Individuals with dietary needs incompatible with the IRCD meal plan
* Individuals with liver or kidney disorders that may be affected by very low glucose and protein content of the diet
* Patients on a calorie restricted diet will also be excluded
* Patients with relevant prior gastrointestinal surgery and consequences such as short bowel syndrome, ostomy of small or large intestine,total colectomy, proctocolectomy, ileoanal pouch will be excluded (not excluded are patients with resection of terminal ileum, resection of short strictures of the small intestine, hemicolectomy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Clinical response as per CDAI (70 points) | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as reduction of the CDAI of at least 70 points or achieving a CDAI score ≤ 150.

SECONDARY OUTCOMES:
Number of Participants with Clinical remission as per CDAI | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as a CDAI score ≤ 150.
Number of Participants with Clinical response as per CDAI (100 points) | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as reduction of the CDAI of at least 100 points or achieving a CDAI score ≤ 150.
Number of Participants with Clinical response as per CDAI (70 points) | Assessed 3 months after 3rd cycle. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as reduction of the CDAI of at least 70 points or achieving a CDAI score ≤ 150.
Change in C-reactive protein (CRP) at baseline versus after 3rd cycle of IRCD (or control at corresponding time point) in both IRCD and control group. | Baseline versus within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Change of the inflammatory marker CRP.
Change in Erythrocyte Sedimentation Rate (ESR) at baseline versus after 3rd cycle of IRCD (or control at corresponding time point) in both IRCD and control group. | Baseline versus within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Change of the inflammatory marker ESR.
Change in fecal calprotectin at baseline versus after 3rd cycle of IRCD (or control at corresponding time point) in both IRCD and control group. | Baseline versus within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Change of the inflammatory marker fecal calprotectin.
Number of Participants with Clinical remission as per Patient Reported Outcome (PRO) score | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as average worst daily abdominal pain score of ≤ 1 (using a 4-point scale, 0-3) and a loose/watery stool (Bristol Type 6 or 7) frequency score of <=3.
Patient global assessment | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  "Do you believe you are in remission from your CD symptoms?" (Yes/No). No scale.
Effect of IRCD on endoscopic outcomes | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Changes in Simplified Endoscopic Activity Score for Crohn's Disease (SES-CD). SES-CD scores range from 0 to 56 and higher scores indicate more severe disease.
Effect of IRCD on patient quality of life: Short Inflammatory Bowel Disease questionnaire (SIBDQ) | Assessed within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Changes in SIBDQ. Response to each of the questions is graded from 1 to 7 (1 being the worst situation and 7 the best).

OTHER OUTCOMES:
Number of Participants with Clinical remission as per CDAI | Assessed 3 months after 3rd cycle. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as a CDAI score ≤ 150.
Number of Participants with Clinical response as per CDAI (100 points) | Assessed 3 months after 3rd cycle. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Defined as reduction of the CDAI of at least 100 points or achieving a CDAI score ≤ 150.
Changes in clinical markers of disease activity | At baseline versus 3 months after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Clinical markers of disease activity are CRP, ESR, and fecal calprotectin.
Effect of IRCD on patient quality of life: Short Inflammatory Bowel Disease questionnaire (SIBDQ) | Assessed 3 months after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Changes in SIBDQ. Response to each of the questions is graded from 1 to 7 (1 being the worst situation and 7 the best).
Changes in clinical markers of disease activity | At baseline versus within 6 days after 1st cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Clinical markers of disease activity are CRP, ESR, and fecal calprotectin.
Changes in cytokines/chemokines and immune cell profiles | At baseline versus within 6 days after 3rd cycle of IRCD. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Using flow cytometry and mass cytometry (CyTOF)
Changes in gut metabolites (including short-chain fatty acid and bile acid profiles) and microbiome profiles (using 16S rRNA/shotgun metagenomics) | At baseline versus within 6 days after 3rd cycle of IRCD and 3 months after 3rd cycle. 1 cycle of IRCD lasts 5 days and is administered once a month, followed by regular diet for the rest of the month.
  Gut metabolites include short-chain fatty acid and bile acid profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha R Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulkarni C, Fardeen T, Gubatan J, Ye J, Jarr K, Dickson E, Jang H, Temby M, Patel A, Jiang Y, Singh G, Keyashian K, Streett S, Ho E, Barber G, Singh S, Limsui D, Anaizi N, Becker L, Spencer SP, Mehrish D, Perelman D, Longo VD, Charu V, Ashouri JF, Davis MM, Habtezion A, Sonnenburg JL, Gardner C, Sinha SR. A fasting-mimicking diet in patients with mild-to-moderate Crohn's disease: a randomized controlled trial. Nat Med. 2026 Jan 13. doi: 10.1038/s41591-025-04173-w. Online ahead of print. PMID 41530382